CLINICAL TRIAL: NCT01429779
Title: The Orange-III Trial: Optimised Recovery With Movicol® Preoperatively Within an Enhanced Recovery Programme, a Randomised Controlled Trial
Brief Title: The Orange-III Trial: Optimised Recovery With Movicol® Preoperatively Within an Enhanced Recovery Programme
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Norgine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 11-1-039
Record Dates: First submitted 2011-09-06; First posted 2011-09-07 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: Liver Diseases
Keywords: General surgery
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Movicol (Experimental): Administration of 1 sachet of Movicol® daily during one week preoperatively (experimental care) and 2 sachets of Movicol® daily postoperatively (standard care).
  Interventions: Drug: Movicol
- Control (No Intervention): Control group; standard postoperative care (administration of 2 sachets of Movicol® postoperatively daily)

INTERVENTIONS:
Drug: Movicol — Movicol® in sachets of 13,81 gram each. One sachet consists of 13,125 gr Macrogol 3350, 178,5 mg Sodium bicarbonate, 350,7 mg Sodium chloride and 46,6 mg Potassium chloride. Administration of 1 sachet of Movicol® daily during one week preoperatively and 2 sachets of Movicol® daily postoperatively.
  Arms: Movicol

SUMMARY:
The aim of this study is to accelerate recovery after liver surgery by enhancing intestinal passage through the preoperative use of Movicol.

Hypothesis The use of Movicol® during one week prior to partial liver resection combined with the Enhanced Recovery After Surgery (ERAS®) programme accelerates functional recovery by promoting early return of gastro-intestinal function, defined as the passage of stools and early oral intake.

DETAILED DESCRIPTION:
Rationale:

The routine use of laxatives after liver surgery as part of an Enhanced Recovery After Surgery (ERAS®) programme enhances recovery of gastro-intestinal function and early tolerance of oral nutrition. The use of Macrogol (Movicol®) as laxative during one week prior to partial liver resection will further enhance early return of gastro-intestinal function and accelerate functional recovery.

Objective:

The aim of this study is to accelerate recovery after liver surgery by enhancing intestinal passage through the preoperative use of Movicol®

Study design:

The Orange-III trial is a multicentre randomised controlled trial to aim whether the administration of 1 sachet of Movicol® during one week preoperatively and 2 sachets of Movicol® postoperatively will further enhance early recovery compared to the administration of 2 sachets of Movicol® postoperatively only, following liver surgery. All patients will be managed within an ERAS® programme of perioperative care.

Study population:

Patients requiring a partial liver resection (two or more segments), 18-80 yr old.

Main study parameters/endpoints:

The main objective of the Orange-III trial is to provide evidence on early recovery of gastro-intestinal function defined as time to first intake of solid food continued for more than 24 hours after the use of Movicol® during one week prior to partial liver resection within an enhanced recovery programme. Secondary objectives are recovery of gastro-intestinal function defined as time to first stools and time to continuous intake of clear fluids for more than 24 hours, functional recovery, hospital length of stay and patient activity level.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a partial liver resection
* Able to understand the nature of the study and what will be required of them
* Men and non-pregnant, non-lactating women between age 18-80
* BMI between 18-35
* Patients with ASA I-III

Exclusion Criteria:

* Inability to give written informed consent
* Patients requiring bile duct reconstruction
* Patients with ASA IV-V
* Superextended hepatectomy
* Underlying symptomatic liver disease such as cirrhosis
* Underlying gastro-intestinal disease such as motility disorders
* Need for procedures additive to partial liver resection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Recovery of gastro-intestinal function | 20 days
  Recovery of gastro-intestinal function defined as time to first intake of solid food continued for more than 24 hours

SECONDARY OUTCOMES:
Recovery of gastro-intestinal function | 20 days
  Recovery of gastro-intestinal function defined as time to continuous oral intake of clear liquids for more than 24 hours
Functional recovery | 20 days
  Functional recovery (measured by the following functional recovery criteria)
  * Adequate pain control on oral analgesics only
  * Eating and drinking properly without the need of IV fluids
  * Independently mobile or mobile at preoperative level
  * Standard laboratory tests and liver function returning to normal level
Hospital length of stay | 20 days

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M van Dam, MD, Principal Investigator — Maastricht University Hospital; Cornelis H.C. Dejong, MD PHD, Study Director — Maastricht University Hospital
Locations (2):
- Universitatsklinikum Aachen, Aachen, Germany
- Maastricht University Hospital, Maastricht, Limburg, Netherlands